CLINICAL TRIAL: NCT01270815
Title: An Open-Label, Single-Dose, Randomized, Four-Way Crossover Study In Healthy Volunteers To Investigate The Pharmacokinetics Of Pregabalin Controlled Release Formulation Administered At Lunch Following Various Caloric Intakes As Compared To The Immediate Release Formulation
Brief Title: An Investigation Of The Absorption And Pharmacokinetics Of A Single Dose Of A Controlled Release (CR) Pregabalin Tablet Following Various Sized Lunches As Compared To A Single Dose Of The Immediate Release (IR) Pregabalin Capsule In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A0081188
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2011-05

CONDITIONS: Healthy
Keywords: pregabalin; pharmacokinetics; bioavailability; bioequivalence
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pregabalin controlled release, 330 mg, 400 to 500 calories (Experimental)
  Interventions: Drug: Pregabalin controlled release, 330 mg, 400 to 500 calories
- Pregabalin controlled release, 330 mg, 600 to 750 calories (Experimental)
  Interventions: Drug: Pregabalin controlled release, 330 mg, 600 to 750 calories
- Pregabalin controlled release, 330 mg, 800 to 1000 calories (Experimental)
  Interventions: Drug: Pregabalin controlled release, 330 mg, 800 to 1000 calories
- Pregabalin immediate release, 300 mg (Other): Reference
  Interventions: Drug: Pregabalin immediate release, 300 mg

INTERVENTIONS:
Drug: Pregabalin controlled release, 330 mg, 400 to 500 calories — A single oral dose of 330 mg controlled release tablet administered following a 400 to 500 calorie medium-fat lunch
  Arms: Pregabalin controlled release, 330 mg, 400 to 500 calories
Drug: Pregabalin controlled release, 330 mg, 600 to 750 calories — A single oral dose of 330 mg controlled release tablet administered following a 600 to 750 calorie medium-fat lunch
  Arms: Pregabalin controlled release, 330 mg, 600 to 750 calories
Drug: Pregabalin controlled release, 330 mg, 800 to 1000 calories — A single oral dose of 330 mg controlled release tablet administered following an 800 to 1000 calorie medium-fat lunch
  Arms: Pregabalin controlled release, 330 mg, 800 to 1000 calories
Drug: Pregabalin immediate release, 300 mg — A single oral dose of 300 mg immediate release capsule administered fasted
  Arms: Pregabalin immediate release, 300 mg

SUMMARY:
The purpose of this study is to 1) evaluate the extent of absorption of a single dose of a pregabalin controlled release tablet following a 400 to 500 calorie, 600 to 750 calorie, or 800 to 1000 calorie medium-fat lunch as compared to pregabalin immediate release capsule 2) evaluate the safety and tolerability of a single dose of a pregabalin controlled release tablet following various sized lunches as compared to a single dose of the pregabalin immediate release capsule.

DETAILED DESCRIPTION:
Evaluate the absorption, pharmacokinetics, safety/tolerability of a single dose of a pregabalin CR tablet under various conditions as compared to single dose of pregabalin IR capsule

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females
* Between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2

Exclusion Criteria:

* Illicit drug use
* Pregnant or nursing females
* Females of childbearing potential who are unwilling or unable to use an acceptable method of contraception

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve from 0 to infinity (AUCinf) for assessment of equivalence between the controlled release treatments and the immediate release treatments | 3 days

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Chew ML, Plotka A, Alvey CW, Pitman VW, Alebic-Kolbah T, Scavone JM, Bockbrader HN. Pharmacokinetics of pregabalin controlled-release in healthy volunteers: effect of food in five single-dose, randomized, clinical pharmacology studies. Clin Drug Investig. 2014 Sep;34(9):617-26. doi: 10.1007/s40261-014-0211-4. PMID 25078976
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081188&StudyName=An%20Investigation%20Of%20The%20Absorption%20And%20Pharmacokinetics%20Of%20A%20Single%20Dose%20Of%20A%20Controlled%20Release%20%28CR%29%20Pregabalin%20Tablet%20Following%20Va